CLINICAL TRIAL: NCT04789577
Title: A Phase I/II Observer-blind, Randomized, Placebo-controlled, Multi-center Trial to Evaluate the Safety and Immunogenicity of Different Formulations of Monovalent Influenza A/Hong Kong/125/2017-like (H7N9) Virus Vaccine With AS03 Adjuvant System, Given as a Two-dose Series to Adults 18 to 64 Years of Age and 65 Years of Age and Older
Brief Title: A Study to Evaluate the Safety and Immunogenicity of GlaxoSmithKline Biologicals' Influenza Vaccine GSK3206641A Administered in Adults 18 to 64 Years of Age and 65 Years of Age and Older
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 209671
Record Dates: First submitted 2021-03-05; First posted 2021-03-09 (Actual); Results first posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-09

CONDITIONS: Influenza, Human
MeSH Terms: conditions — Influenza, Human | interventions — AS03 adjuvant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- FLU-Q-PAN H7N9 Formulation 1_B Group (Active Comparator): Healthy male and female participants who received two doses of FLU-Q-PAN H7N9 Formulation 1 vaccine and AS03B adjuvant. Participants received the first dose at Day 1 and the second dose at Day 22.
  Interventions: Biological: FLU-Q-PAN H7N9 Formulation 1; Biological: AS03B
- FLU-Q-PAN H7N9 Formulation 1_A Group (Active Comparator): Healthy male and female participants who received two doses of FLU-Q-PAN H7N9 Formulation 1 vaccine and AS03A adjuvant. Participants received the first dose at Day 1 and the second dose at Day 22.
  Interventions: Biological: FLU-Q-PAN H7N9 Formulation 1; Biological: AS03A
- FLU-Q-PAN H7N9 Formulation 2_B Group (Active Comparator): Healthy male and female participants who received two doses of FLU-Q-PAN H7N9 Formulation 2 vaccine and AS03B adjuvant. Participants received the first dose at Day 1 and the second dose at Day 22.
  Interventions: Biological: FLU-Q-PAN H7N9 Formulation 2; Biological: AS03B
- FLU-Q-PAN H7N9 Formulation 2_A Group (Active Comparator): Healthy male and female participants who received two doses of FLU-Q-PAN H7N9 Formulation 2 vaccine and AS03A adjuvant. Participants received the first dose at Day 1 and the second dose at Day 22.
  Interventions: Biological: FLU-Q-PAN H7N9 Formulation 2; Biological: AS03A
- FLU-Q-PAN H7N9 Formulation 3_B Group (Active Comparator): Healthy male and female participants who received two doses of FLU-Q-PAN H7N9 Formulation 3 vaccine and AS03B adjuvant. Participants received the first dose at Day 1 and the second dose at Day 22.
  Interventions: Biological: FLU-Q-PAN H7N9 Formulation 3; Biological: AS03B
- FLU-Q-PAN H7N9 Formulation 3_A Group (Active Comparator): Healthy male and female participants who received two doses of FLU-Q-PAN H7N9 Formulation 3 vaccine and AS03A adjuvant. Participants received the first dose at Day 1 and the second dose at Day 22.
  Interventions: Biological: FLU-Q-PAN H7N9 Formulation 3; Biological: AS03A
- Placebo Group (Placebo Comparator): Healthy male and female participants who received two doses of placebo, the first dose at Day 1 and the second dose at Day 22.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: FLU-Q-PAN H7N9 Formulation 1 — Participants received two doses of the FLU-Q-PAN H7N9 Formulation 1 vaccine by intramuscular injection in the non-dominant arm.
  Arms: FLU-Q-PAN H7N9 Formulation 1_A Group; FLU-Q-PAN H7N9 Formulation 1_B Group
Biological: FLU-Q-PAN H7N9 Formulation 2 — Participants received two doses of the FLU-Q-PAN H7N9 Formulation 2 vaccine by intramuscular injection in the non-dominant arm.
  Arms: FLU-Q-PAN H7N9 Formulation 2_A Group; FLU-Q-PAN H7N9 Formulation 2_B Group
Biological: FLU-Q-PAN H7N9 Formulation 3 — Participants received two doses of the FLU-Q-PAN H7N9 Formulation 3 vaccine by intramuscular injection in the non-dominant arm.
  Arms: FLU-Q-PAN H7N9 Formulation 3_A Group; FLU-Q-PAN H7N9 Formulation 3_B Group
Biological: AS03B — Participants received two doses of the AS03B adjuvant by intramuscular injection in the non-dominant arm.
  Arms: FLU-Q-PAN H7N9 Formulation 1_B Group; FLU-Q-PAN H7N9 Formulation 2_B Group; FLU-Q-PAN H7N9 Formulation 3_B Group
Biological: AS03A — Participants received two doses of the AS03A adjuvant by intramuscular injection in the non-dominant arm.
  Arms: FLU-Q-PAN H7N9 Formulation 1_A Group; FLU-Q-PAN H7N9 Formulation 2_A Group; FLU-Q-PAN H7N9 Formulation 3_A Group
Drug: Placebo — Participants received two doses of Placebo by intramuscular injection in the non-dominant arm.
  Arms: Placebo Group

SUMMARY:
Study to evaluate the safety and immunogenicity of H7N9 antigen in combination with full or half doses of AS03 adjuvant system in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants as established by medical history and clinical examination before entering into the study.
* A male or female ≥ 18 years of age at the time of first vaccination.
* Participants, who, in the opinion of the investigator, can and will comply with the requirements of the protocol (e.g. completion of the diary cards and COVID-19 assessment card, return for follow-up visits, or return the diary cards and COVID-19 assessment card in a timely manner using the pre stamped envelope received at the site).
* Written or witnessed/thumb printed informed consent obtained from the participant prior to performance of any study specific procedure.
* Female participants of non-childbearing potential may be enrolled in the study. Non childbearing potential is defined as pre-menarche, current bilateral tubal ligation or occlusion hysterectomy, bilateral ovariectomy or post-menopause.
* Female participants of childbearing potential may be enrolled in the study, if the participant:

  * has practiced adequate contraception for 1 month prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Current diagnosis or history of autoimmune disorder(s).
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine.
* Hypersensitivity to latex.
* Acute or chronic clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality that appears uncontrolled, as determined by history or physical examination.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* Recurrent history or uncontrolled neurological disorders or seizures.
* History of Guillain-Barré syndrome.
* Diagnosed with narcolepsy; or history of narcolepsy in a participant's parent, sibling or child.
* Diagnosed with cancer, or treatment for cancer within 3 years.
* Persons with a history of cancer who are disease-free without treatment for 3 years or more are eligible.
* Persons with a history of histologically-confirmed basal cell carcinoma of the skin successfully treated with local excision only are accepted and are eligible, but other histologic types of skin cancer are exclusionary.
* Women who are disease-free 3 years or more after treatment for breast cancer and receiving long-term prophylaxis (for example, with tamoxifen) are eligible.
* Documented human immunodeficiency virus-positive participant.
* Any clinically significant* hematological laboratory abnormality.

  *The investigator should use his/her clinical judgement to decide which abnormalities are clinically significant.
* Bedridden participants.
* Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the participant due to participation in the study.
* Use of any investigational or non-registered product (drug, vaccine or medical device) other than the study vaccine/product during the period beginning 30 days before the first dose of study vaccine/product (Day -29 to Day 1), or planned use during the study period.
* Administration of long-acting immune-modifying drugs at any time during the study period (e.g. infliximab).
* Administration of immunoglobulins and/or any blood products or plasma derivatives during the period starting 3 months before the first dose of study vaccine/product or planned administration during the study period.
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs during the period starting 3 months prior to the first vaccine/product dose. For corticosteroids, this will mean prednisone equivalent ≥ 20 mg/day. Inhaled and topical steroids are allowed.
* Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational vaccine/product (drug or medical device).
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions within 2 months after completion of the vaccination series.
* History of or current chronic alcohol consumption and/or drug abuse.
* Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the participant due to participation in the study.
* Any study personnel or immediate dependents, family, or household member.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 833 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2022-09-12 (Actual); Study Completion 2022-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- United States (8):
  - GSK Investigational Site, Stockbridge, Georgia
  - GSK Investigational Site, Meridian, Idaho
  - GSK Investigational Site, Cary, North Carolina
  - GSK Investigational Site, Wilmington, North Carolina
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Mt. Pleasant, South Carolina
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, West Jordan, Utah

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.

REFERENCES:
- [Derived] Hastie A, Clarke T, Germain S, Ollinger T, Lese P, Gupta V. Immunogenicity and Safety of AS03-Adjuvanted H7N9 Influenza Vaccine in Adults (18-64 and >/=65 Years): A Phase 1/2, Randomized, Placebo-Controlled Trial. Influenza Other Respir Viruses. 2024 Dec;18(12):e70020. doi: 10.1111/irv.70020. PMID 39702896

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Group: Healthy male and female participants who will receive two doses of placebo, the first dose at Day 1 and the second dose at Day 22.
Period: Overall Study
Arm/Group | FLU-Q-PAN H7N9 Formulation 1_B Group | FLU-Q-PAN H7N9 Formulation 1_A Group | FLU-Q-PAN H7N9 Formulation 2_B Group | FLU-Q-PAN H7N9 Formulation 2_A Group | FLU-Q-PAN H7N9 Formulation 3_B Group | FLU-Q-PAN H7N9 Formulation 3_A Group | Placebo Group
Started | 121 | 116 | 119 | 119 | 117 | 121 | 120
Completed | 113 | 103 | 111 | 105 | 108 | 107 | 109
Not Completed | 8 | 13 | 8 | 14 | 9 | 14 | 11
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 3 | 1 | 7 | 1
Not completed — Lost to Follow-up | 7 | 12 | 7 | 10 | 8 | 6 | 10
Not completed — Migrated Or Moved From The Study Area | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — AE Requiring Expedited Reporting | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FLU-Q-PAN H7N9 Formulation 1_B Group | FLU-Q-PAN H7N9 Formulation 1_A Group | FLU-Q-PAN H7N9 Formulation 2_B Group | FLU-Q-PAN H7N9 Formulation 2_A Group | FLU-Q-PAN H7N9 Formulation 3_B Group | FLU-Q-PAN H7N9 Formulation 3_A Group | Placebo Group | Total
Number analyzed (Participants) | 121 | 116 | 119 | 119 | 117 | 121 | 120 | 833
Age, Customized [Count of Participants; unit: Participants]
  18 - 64 years | 61 | 56 | 59 | 59 | 58 | 61 | 60 | 414
  ≥65 years | 60 | 60 | 60 | 60 | 59 | 60 | 60 | 419
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 65 | 74 | 69 | 74 | 67 | 72 | 489
  Male | 53 | 51 | 45 | 50 | 43 | 54 | 48 | 344
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 7 | 14 | 7 | 11 | 5 | 4 | 56
  Not Hispanic or Latino | 113 | 109 | 105 | 112 | 106 | 116 | 116 | 777
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 2 | 2 | 1 | 5 | 2 | 14
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 21 | 19 | 14 | 13 | 19 | 22 | 21 | 129
  White | 98 | 95 | 102 | 104 | 97 | 94 | 96 | 686
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Seroprotected Participants for Anti-hemagglutination Inhibition (HI) Antibodies Against Vaccine-homologous H7N9
Description: Center for Biologics Evaluation and Research (CBER) criteria for seroprotection rate (SPR) for 18 to 64 years of age is shown if the Lower Limit (LL) of the 99.17% confidence interval (CI) for the SPR meets or exceeds 70%, and for greater than or equal to (≥) 65 years of age if the LL of the 99.17% CI for the SPR meets or exceeds 60%. SPR is defined as the percentage of participants with an HI antibody titer ≥40 1/dilution (DIL). The percentage of participants was calculated along with Clopper-Pearson exact two-sided 99.17% CIs.
Time Frame: At Day 43
Population: Analysis was performed on the Per Protocol Set (PPS), which included all participants with no major protocol deviations that lead to exclusion at or prior to Day 43, who had data collected for anti-HI antibodies, at each visit and for whom post-vaccination immunogenicity data was available at Day 43.
Measure: Number (99.17% Confidence Interval); unit: Percentage of Participants
Arm/Group | FLU-Q-PAN H7N9 Formulation 1_B Group | FLU-Q-PAN H7N9 Formulation 1_A Group | FLU-Q-PAN H7N9 Formulation 2_B Group | FLU-Q-PAN H7N9 Formulation 2_A Group | FLU-Q-PAN H7N9 Formulation 3_B Group | FLU-Q-PAN H7N9 Formulation 3_A Group | Placebo Group
Number analyzed (Participants) | 98 | 93 | 97 | 94 | 101 | 94 | 95
Percentage of Participants | 27.1 [16.1 to 40.6] | 27.7 [15.8 to 42.4] | 23.5 [12.7 to 37.6] | 26.5 [14.9 to 41.1] | 19.1 [9.5 to 32.3] | 40.5 [26.7 to 55.4] | 0 [0 to 0]

2. Primary Outcome: Percentage of Seroconverted Participants for Anti-HI Antibodies Against Vaccine-homologous H7N9
Description: CBER criteria for seroconversion rate (SCR) for 18 to 64 years of age is shown if LL of the 99.17% CI for the SCR meets or exceeds 40%, and for ≥65 years of age, if the LL of the 99.17% CI for the SCR meets or exceeds 30%. Seroconversion is defined as a post-vaccination antibody titer ≥40 1/DIL in the serum of participants seronegative before vaccination (i.e. titer < assay cut-off at Day 1). For seropositive participants (i.e. titer ≥ assay cut-off at Day 1), seroconversion requires a 4-fold rise in post-vaccination HI antibody titer (but at least a titer of 40 1/DIL). The percentage of participants was calculated with Clopper-Pearson exact two-sided 99.17% CIs.
  Note: The cut-off value for antibody titer was defined by the laboratory before the analysis.
Time Frame: At Day 43
Population: as for outcome 1
Measure: Number (99.17% Confidence Interval); unit: Percentage of Participants
Arm/Group | FLU-Q-PAN H7N9 Formulation 1_B Group | FLU-Q-PAN H7N9 Formulation 1_A Group | FLU-Q-PAN H7N9 Formulation 2_B Group | FLU-Q-PAN H7N9 Formulation 2_A Group | FLU-Q-PAN H7N9 Formulation 3_B Group | FLU-Q-PAN H7N9 Formulation 3_A Group | Placebo Group
Number analyzed (Participants) | 98 | 93 | 97 | 94 | 101 | 94 | 95
Percentage of Participants | 27.1 [16.1 to 40.6] | 27.7 [15.8 to 42.4] | 23.5 [12.7 to 37.6] | 26.5 [14.9 to 41.1] | 19.1 [9.5 to 32.3] | 40.5 [26.7 to 55.4] | 0 [0 to 0]

3. Primary Outcome: Number of Participants With Any Solicited Administration Site Events
Description: Solicited administered site events assessed were pain, redness and swelling. Any Pain = occurrence of symptom regardless of intensity grade. Any Redness or any Swelling symptom = any symptom having a surface diameter greater than (>) 20 millimeters (mm).
Time Frame: Within the 7-day follow-up period after Dose 1
Population: Analysis was performed on the Exposed Set, which included all participants who received the first dose of study intervention and had solicited administration site adverse events data.
Measure: Count of Participants; unit: Participants
Arm/Group | FLU-Q-PAN H7N9 Formulation 1_B Group | FLU-Q-PAN H7N9 Formulation 1_A Group | FLU-Q-PAN H7N9 Formulation 2_B Group | FLU-Q-PAN H7N9 Formulation 2_A Group | FLU-Q-PAN H7N9 Formulation 3_B Group | FLU-Q-PAN H7N9 Formulation 3_A Group | Placebo Group
Number analyzed (Participants) | 121 | 113 | 117 | 117 | 114 | 115 | 118
Participants
  Any Pain | 72 | 77 | 68 | 80 | 53 | 78 | 15
  Any Redness | 1 | 3 | 2 | 5 | 0 | 2 | 0
  Any Swelling | 1 | 6 | 4 | 5 | 0 | 2 | 0

4. Primary Outcome: Number of Participants With Any Solicited Administration Site Events
Description: Solicited administered site events assessed were pain, redness and swelling. Any Pain = occurrence of symptom regardless of intensity grade. Any Redness or any Swelling symptom = any symptom having a surface diameter >20 mm.
Time Frame: Within the 7-day follow-up period after Dose 2
Population: Analysis was performed on the Exposed Set, which included all participants who received the second dose of study intervention and had solicited administration site adverse events data.
Measure: Count of Participants; unit: Participants
Arm/Group | FLU-Q-PAN H7N9 Formulation 1_B Group | FLU-Q-PAN H7N9 Formulation 1_A Group | FLU-Q-PAN H7N9 Formulation 2_B Group | FLU-Q-PAN H7N9 Formulation 2_A Group | FLU-Q-PAN H7N9 Formulation 3_B Group | FLU-Q-PAN H7N9 Formulation 3_A Group | Placebo Group
Number analyzed (Participants) | 112 | 107 | 112 | 108 | 106 | 105 | 111
Participants
  Any Pain | 53 | 62 | 58 | 66 | 42 | 56 | 13
  Any Redness | 1 | 3 | 0 | 3 | 1 | 2 | 0
  Any Swelling | 4 | 8 | 1 | 5 | 1 | 4 | 0

5. Primary Outcome: Number of Participants With Any Solicited Systemic Events
Description: Solicited systemic events assessed were fatigue, fever, headache, muscle ache all over body, joint pain, shivering, sweating and gastrointestinal symptoms (Nausea, vomiting, diarrhea and abdominal pain). Any = occurrence of symptom regardless of intensity grade. Fever was defined as temperature ≥38 degrees Celsius (°C) for oral route (preferred location for measuring temperature).
Time Frame: Within the 7-day follow-up period after Dose 1
Population: Analysis was performed on the Exposed Set, which included all participants who received the first dose of study intervention and had solicited systemic adverse events data.
Measure: Count of Participants; unit: Participants
Arm/Group | FLU-Q-PAN H7N9 Formulation 1_B Group | FLU-Q-PAN H7N9 Formulation 1_A Group | FLU-Q-PAN H7N9 Formulation 2_B Group | FLU-Q-PAN H7N9 Formulation 2_A Group | FLU-Q-PAN H7N9 Formulation 3_B Group | FLU-Q-PAN H7N9 Formulation 3_A Group | Placebo Group
Number analyzed (Participants) | 121 | 112 | 117 | 117 | 114 | 115 | 118
Participants
  Any Fatigue | 41 | 39 | 31 | 36 | 27 | 41 | 37
  Any Fever | 2 | 1 | 1 | 1 | 0 | 2 | 0
  Any Headache | 31 | 29 | 24 | 33 | 16 | 33 | 29
  Any Muscle Ache (all over body) | 27 | 20 | 16 | 21 | 12 | 25 | 8
  Any Joint Pain | 13 | 13 | 19 | 11 | 12 | 16 | 10
  Any Shivering | 7 | 6 | 8 | 4 | 5 | 8 | 6
  Any Sweating | 10 | 7 | 4 | 4 | 7 | 13 | 8
  Any Nausea | 9 | 9 | 11 | 11 | 8 | 8 | 5
  Any Vomiting | 2 | 1 | 2 | 2 | 0 | 1 | 0
  Any Diarrhea | 7 | 10 | 15 | 8 | 6 | 8 | 11
  Any Abdominal Pain | 5 | 9 | 7 | 6 | 6 | 8 | 3

6. Primary Outcome: Number of Participants With Any Solicited Systemic Events
Description: Solicited systemic events assessed were fatigue, fever, headache, muscle ache all over body, joint pain, shivering, sweating and gastrointestinal symptoms (Nausea, vomiting, diarrhea and abdominal pain). Any = occurrence of symptom regardless of intensity grade. Fever was defined as temperature ≥38°C for oral route (preferred location for measuring temperature).
Time Frame: Within the 7-day follow-up period after Dose 2
Population: Analysis was performed on the Exposed Set, which included all participants who received the second dose of study intervention and had solicited systemic adverse events data.
Measure: Count of Participants; unit: Participants
Arm/Group | FLU-Q-PAN H7N9 Formulation 1_B Group | FLU-Q-PAN H7N9 Formulation 1_A Group | FLU-Q-PAN H7N9 Formulation 2_B Group | FLU-Q-PAN H7N9 Formulation 2_A Group | FLU-Q-PAN H7N9 Formulation 3_B Group | FLU-Q-PAN H7N9 Formulation 3_A Group | Placebo Group
Number analyzed (Participants) | 112 | 107 | 112 | 108 | 106 | 105 | 111
Participants
  Any Fatigue | 34 | 20 | 28 | 29 | 21 | 34 | 20
  Any Fever | 1 | 2 | 0 | 3 | 0 | 2 | 0
  Any Headache | 23 | 19 | 19 | 20 | 16 | 21 | 12
  Any Muscle Ache (all over body) | 14 | 14 | 18 | 15 | 9 | 16 | 2
  Any Joint Pain | 8 | 10 | 15 | 12 | 10 | 14 | 6
  Any Shivering | 9 | 4 | 6 | 3 | 2 | 6 | 1
  Any Sweating | 6 | 4 | 7 | 7 | 6 | 8 | 5
  Any Nausea | 6 | 8 | 10 | 6 | 7 | 7 | 5
  Any Vomiting | 1 | 5 | 0 | 1 | 0 | 0 | 1
  Any Diarrhea | 5 | 5 | 9 | 7 | 6 | 4 | 7
  Any Abdominal Pain | 5 | 1 | 10 | 5 | 5 | 5 | 5

7. Primary Outcome: Number of Participants With Any and Related Unsolicited Adverse Events
Description: An unsolicited adverse event (AE) is an AE that was not solicited using a Participant Diary and that was spontaneously communicated by a participant who had signed the informed consent. Unsolicited AEs include serious and non-serious AEs. Potential unsolicited AEs may have been medically attended (i.e. symptoms or illnesses requiring a hospitalization, or emergency room visit, or visit to/by a health care provider). Unsolicited AEs that were not medically attended nor perceived as a concern by participant were collected during interview with the participants and by review of available medical records at the following visit. An unsolicited adverse event is any event reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: Within the 21-day follow-up period after Dose 1
Population: Analysis was performed on the ES, which included all participants who received the first dose of study intervention and had unsolicited adverse events data.
Measure: Count of Participants; unit: Participants
Arm/Group | FLU-Q-PAN H7N9 Formulation 1_B Group | FLU-Q-PAN H7N9 Formulation 1_A Group | FLU-Q-PAN H7N9 Formulation 2_B Group | FLU-Q-PAN H7N9 Formulation 2_A Group | FLU-Q-PAN H7N9 Formulation 3_B Group | FLU-Q-PAN H7N9 Formulation 3_A Group | Placebo Group
Number analyzed (Participants) | 121 | 116 | 119 | 119 | 117 | 121 | 120
Participants
  Any AEs | 26 | 19 | 20 | 21 | 15 | 26 | 21
  Related AEs | 9 | 7 | 7 | 10 | 9 | 13 | 8

8. Primary Outcome: Number of Participants With Any and Related Unsolicited Adverse Events
Description: An unsolicited AE is an AE that was not solicited using a Participant Diary and that was spontaneously communicated by a participant who has signed the informed consent. Unsolicited AEs include serious and non-serious AEs. Potential unsolicited AEs may have been medically attended (i.e. symptoms or illnesses requiring a hospitalization, or emergency room visit, or visit to/by a health care provider). Unsolicited AEs that were not medically attended nor perceived as a concern by participant are collected during interview with the participants and by review of available medical records at the next visit. An unsolicited adverse event is any event reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: Within the 21-day follow-up period after Dose 2
Population: Analysis was performed on the ES, which included all participants who received the second dose of study intervention and had unsolicited adverse events data.
Measure: Count of Participants; unit: Participants
Arm/Group | FLU-Q-PAN H7N9 Formulation 1_B Group | FLU-Q-PAN H7N9 Formulation 1_A Group | FLU-Q-PAN H7N9 Formulation 2_B Group | FLU-Q-PAN H7N9 Formulation 2_A Group | FLU-Q-PAN H7N9 Formulation 3_B Group | FLU-Q-PAN H7N9 Formulation 3_A Group | Placebo Group
Number analyzed (Participants) | 115 | 112 | 113 | 111 | 111 | 106 | 113
Participants
  Any AEs | 20 | 20 | 16 | 19 | 19 | 21 | 14
  Related AEs | 4 | 7 | 5 | 3 | 8 | 7 | 7

9. Primary Outcome: Number of Participants With Any and Related Medically Attended Adverse Events (MAEs)
Description: MAEs were defined as adverse events with medically-attended visits that are not routine visits for physical examination or vaccination, such as visits for hospitalization, an emergency room visit, or an otherwise unscheduled visit to or from medical personnel (medical doctor) for any reason.
Time Frame: Within the 21-day follow-up period after Dose 1
Population: Analysis was performed on the ES, which included all participants who received the first dose of study intervention and had MAEs data.
Measure: Count of Participants; unit: Participants
Arm/Group | FLU-Q-PAN H7N9 Formulation 1_B Group | FLU-Q-PAN H7N9 Formulation 1_A Group | FLU-Q-PAN H7N9 Formulation 2_B Group | FLU-Q-PAN H7N9 Formulation 2_A Group | FLU-Q-PAN H7N9 Formulation 3_B Group | FLU-Q-PAN H7N9 Formulation 3_A Group | Placebo Group
Number analyzed (Participants) | 121 | 116 | 119 | 119 | 117 | 121 | 120
Participants
  Any MAEs | 5 | 7 | 10 | 5 | 3 | 9 | 4
  Related MAEs | 1 | 0 | 1 | 0 | 2 | 1 | 0

10. Primary Outcome: Number of Participants With Any and Related MAEs
Description: as for outcome 9
Time Frame: Within the 21-day follow-up period after Dose 2
Population: Analysis was performed on the ES, which included all participants who received the second dose of study intervention and had MAEs data.
Measure: Count of Participants; unit: Participants
Arm/Group | FLU-Q-PAN H7N9 Formulation 1_B Group | FLU-Q-PAN H7N9 Formulation 1_A Group | FLU-Q-PAN H7N9 Formulation 2_B Group | FLU-Q-PAN H7N9 Formulation 2_A Group | FLU-Q-PAN H7N9 Formulation 3_B Group | FLU-Q-PAN H7N9 Formulation 3_A Group | Placebo Group
Number analyzed (Participants) | 115 | 112 | 113 | 111 | 111 | 106 | 113
Participants
  Any MAEs | 6 | 7 | 4 | 8 | 3 | 7 | 3
  Related MAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0

11. Primary Outcome: Number of Participants With Any and Related Serious Adverse Events (SAEs)
Description: A SAE is any untoward medical occurrence that results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization or result in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant. Abnormal pregnancy outcomes were also considered (e.g. spontaneous abortion, fatal death, stillbirth, congenital anomalies, ectopic pregnancy) or other situations where medical or scientific judgement was exercised in deciding whether reporting was appropriate.
Time Frame: From Day 1 up to Day 43
Population: Analysis was performed on the ES, which included all participants who received any study intervention and had SAEs data.
Measure: Count of Participants; unit: Participants
Arm/Group | FLU-Q-PAN H7N9 Formulation 1_B Group | FLU-Q-PAN H7N9 Formulation 1_A Group | FLU-Q-PAN H7N9 Formulation 2_B Group | FLU-Q-PAN H7N9 Formulation 2_A Group | FLU-Q-PAN H7N9 Formulation 3_B Group | FLU-Q-PAN H7N9 Formulation 3_A Group | Placebo Group
Number analyzed (Participants) | 121 | 116 | 119 | 119 | 117 | 121 | 120
Participants
  Any SAEs | 0 | 1 | 1 | 0 | 2 | 0 | 0
  Related SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0

12. Primary Outcome: Number of Participants With Any and Related Potential Immune Mediated Diseases (pIMDs)
Description: pIMDs are a subset of adverse events of special interest that included autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have had an autoimmune etiology.
Time Frame: From Day 1 up to Day 43
Population: Analysis was performed on the ES, which included all participants who received any study intervention and had pIMDs adverse events data.
Measure: Count of Participants; unit: Participants
Arm/Group | FLU-Q-PAN H7N9 Formulation 1_B Group | FLU-Q-PAN H7N9 Formulation 1_A Group | FLU-Q-PAN H7N9 Formulation 2_B Group | FLU-Q-PAN H7N9 Formulation 2_A Group | FLU-Q-PAN H7N9 Formulation 3_B Group | FLU-Q-PAN H7N9 Formulation 3_A Group | Placebo Group
Number analyzed (Participants) | 121 | 116 | 119 | 119 | 117 | 121 | 120
Participants
  Any pIMDs | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related pIMDs | 0 | 0 | 0 | 0 | 0 | 0 | 0

13. Primary Outcome: Number of Participants With Any pIMDs
Description: as for outcome 12
Time Frame: From Day 1 up to Month 13
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | FLU-Q-PAN H7N9 Formulation 1_B Group | FLU-Q-PAN H7N9 Formulation 1_A Group | FLU-Q-PAN H7N9 Formulation 2_B Group | FLU-Q-PAN H7N9 Formulation 2_A Group | FLU-Q-PAN H7N9 Formulation 3_B Group | FLU-Q-PAN H7N9 Formulation 3_A Group | Placebo Group
Number analyzed (Participants) | 121 | 116 | 119 | 119 | 117 | 121 | 120
Participants | 0 | 0 | 1 | 1 | 0 | 2 | 0

14. Primary Outcome: Number of Participants With Any SAEs
Description: as for outcome 11
Time Frame: From Day 1 up to Month 13
Population: Analysis was performed on the ES, which included all participants who received any study intervention and had SAEs data.
Measure: Count of Participants; unit: Participants
Arm/Group | FLU-Q-PAN H7N9 Formulation 1_B Group | FLU-Q-PAN H7N9 Formulation 1_A Group | FLU-Q-PAN H7N9 Formulation 2_B Group | FLU-Q-PAN H7N9 Formulation 2_A Group | FLU-Q-PAN H7N9 Formulation 3_B Group | FLU-Q-PAN H7N9 Formulation 3_A Group | Placebo Group
Number analyzed (Participants) | 121 | 116 | 119 | 119 | 117 | 121 | 120
Participants | 3 | 3 | 10 | 4 | 6 | 5 | 7

15. Secondary Outcome: HI Antibody Titers Against Vaccine-homologous H7N9
Description: HI antibody titers were expressed as Geometric Mean Titers (GMTs). The GMTs calculations were performed by taking the anti-log of the mean of the titer transformations. Values for titers below the assay cutoff will be assigned half the assay cut-off value for the purpose of GMT computation.
  Note: The cut-off value for HI titer was defined by the laboratory before the analysis.
Time Frame: At Day 1, Day 22 and Day 43
Population: Analysis was performed on the PPS, which included all participants with no major protocol deviations that lead to exclusion at or prior to Day 43, who had data collected for HI antibody titers at each visit and for whom post-vaccination immunogenicity data was available for the specified timepoints and specific assay.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | FLU-Q-PAN H7N9 Formulation 1_B Group | FLU-Q-PAN H7N9 Formulation 1_A Group | FLU-Q-PAN H7N9 Formulation 2_B Group | FLU-Q-PAN H7N9 Formulation 2_A Group | FLU-Q-PAN H7N9 Formulation 3_B Group | FLU-Q-PAN H7N9 Formulation 3_A Group | Placebo Group
Number analyzed (Participants) | 98 | 93 | 97 | 94 | 101 | 94 | 95
Titers
  Day 1 | 5.2 [5.0 to 5.4] | 5.2 [5.0 to 5.5] | 5.1 [5.0 to 5.2] | 5.1 [5.0 to 5.2] | 5.1 [5.0 to 5.3] | 5.1 [5.0 to 5.3] | 5.1 [5.0 to 5.2]
  Day 22 | 5.9 [5.4 to 6.4] | 6.0 [5.6 to 6.4] | 6.8 [5.9 to 8.0] | 7.0 [6.2 to 8.0] | 7.6 [6.5 to 8.8] | 8.9 [7.4 to 10.7] | 5.1 [5.0 to 5.2]
  Day 43: number analyzed (Participants) | 96 | 83 | 85 | 83 | 89 | 84 | 82
  Day 43 | 13.8 [11.4 to 16.7] | 15.7 [13.0 to 18.9] | 14.1 [11.4 to 17.3] | 16.4 [13.6 to 19.7] | 13.3 [10.9 to 16.2] | 23.1 [18.2 to 29.3] | 5.1 [5.0 to 5.3]

16. Secondary Outcome: Percentage of Seropositive Participants for HI Antibodies Against Vaccine-homologous H7N9
Description: A seropositive participant is a participant whose antibody titer was greater than or equal to the assay cut-off value.
  Note: The cut-off value for antibody titer was defined by the laboratory before the analysis.
Time Frame: At Day 1, Day 22 and Day 43
Population: Analysis was performed on the PPS, which included all participants with no major protocol deviations that lead to exclusion at or prior to Day 43, who had data collected for anti-HI antibodies, at each visit and for whom post-vaccination immunogenicity data was available for the specified timepoints and specific assay.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | FLU-Q-PAN H7N9 Formulation 1_B Group | FLU-Q-PAN H7N9 Formulation 1_A Group | FLU-Q-PAN H7N9 Formulation 2_B Group | FLU-Q-PAN H7N9 Formulation 2_A Group | FLU-Q-PAN H7N9 Formulation 3_B Group | FLU-Q-PAN H7N9 Formulation 3_A Group | Placebo Group
Number analyzed (Participants) | 98 | 93 | 97 | 94 | 101 | 94 | 95
Percentage of Participants
  Day 1 | 4.1 [1.1 to 10.1] | 4.3 [1.2 to 10.6] | 3.1 [0.6 to 8.8] | 3.2 [0.7 to 9.0] | 2.0 [0.2 to 7.0] | 4.3 [1.2 to 10.5] | 2.1 [0.3 to 7.4]
  Day 22 | 18.4 [11.3 to 27.5] | 24.7 [16.4 to 34.8] | 23.7 [15.7 to 33.4] | 29.8 [20.8 to 40.1] | 32.7 [23.7 to 42.7] | 44.7 [34.4 to 55.3] | 3.2 [0.7 to 9.0]
  Day 43: number analyzed (Participants) | 96 | 83 | 85 | 83 | 89 | 84 | 82
  Day 43 | 65.6 [55.2 to 75.0] | 77.1 [66.6 to 85.6] | 71.8 [61.0 to 81.0] | 79.5 [69.2 to 87.6] | 69.7 [59.0 to 79.0] | 83.3 [73.6 to 90.6] | 3.7 [0.8 to 10.3]

17. Secondary Outcome: Percentage of Seroconverted Participants for HI Antibodies Against Vaccine-homologous H7N9
Description: Seroconversion rate is defined as the percentage of participants with a post-vaccination antibody titer ≥40 1/DIL in the serum of participants seronegative before vaccination (i.e. titer < assay cut-off at Day 1). For seropositive participants (i.e. titer ≥ assay cut-off at Day 1), seroconversion required a 4-fold rise in post-vaccination HI antibody titer (but at least a titer of 40 1/DIL).
  Note: The cut-off value for antibody titer was defined by the laboratory before the analysis.
Time Frame: At Day 22
Population: Analysis was performed on the PPS, which included all participants with no major protocol deviations that lead to exclusion at or prior to Day 22, who had data collected for anti-HI antibodies, at each visit and for whom post-vaccination immunogenicity data was available at Day 22.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | FLU-Q-PAN H7N9 Formulation 1_B Group | FLU-Q-PAN H7N9 Formulation 1_A Group | FLU-Q-PAN H7N9 Formulation 2_B Group | FLU-Q-PAN H7N9 Formulation 2_A Group | FLU-Q-PAN H7N9 Formulation 3_B Group | FLU-Q-PAN H7N9 Formulation 3_A Group | Placebo Group
Number analyzed (Participants) | 98 | 93 | 97 | 94 | 101 | 94 | 95
Percentage of Participants | 0 [0.0 to 3.7] | 0 [0.0 to 3.9] | 5.2 [1.7 to 11.6] | 4.3 [1.2 to 10.5] | 6.9 [2.8 to 13.8] | 9.6 [4.5 to 17.4] | 0 [0.0 to 3.8]

18. Secondary Outcome: Percentage of Seroprotected Participants for HI Antibodies Against Vaccine-homologous H7N9
Description: SPR is defined as the percentage of participants with HI antibody titer ≥40 1/DIL.
  Note: The cut-off value for antibody titer was defined by the laboratory before the analysis.
Time Frame: At Day 1 and Day 22
Population: Analysis was performed on the Per Protocol Set (PPS), which included all participants with no major protocol deviations that lead to exclusion at or prior to Day 22, who had data collected for anti-HI antibodies, at each visit and for whom post-vaccination immunogenicity data was available at the specified timepoints and specific assay.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | FLU-Q-PAN H7N9 Formulation 1_B Group | FLU-Q-PAN H7N9 Formulation 1_A Group | FLU-Q-PAN H7N9 Formulation 2_B Group | FLU-Q-PAN H7N9 Formulation 2_A Group | FLU-Q-PAN H7N9 Formulation 3_B Group | FLU-Q-PAN H7N9 Formulation 3_A Group | Placebo Group
Number analyzed (Participants) | 98 | 93 | 97 | 94 | 101 | 94 | 95
Percentage of Participants
  Day 1 | 0 [0.0 to 3.7] | 1.1 [0.0 to 5.8] | 0 [0.0 to 3.7] | 0 [0.0 to 3.8] | 0 [0.0 to 3.6] | 0 [0.0 to 3.8] | 0 [0.0 to 3.8]
  Day 22 | 1.0 [0.0 to 5.6] | 0 [0.0 to 3.9] | 5.2 [1.7 to 11.6] | 4.3 [1.2 to 10.5] | 6.9 [2.8 to 13.8] | 9.6 [4.5 to 17.4] | 0 [0.0 to 3.8]

19. Secondary Outcome: Mean Geometric Increase (MGI) of HI Antibody Titers Against Vaccine-homologous H7N9
Description: MGI was defined as the fold increase in serum HI GMTs post-vaccination compared to pre-vaccination (Day 1): post-vaccination GMT over pre-vaccination GMT.
Time Frame: At Day 22 (post-Dose 1/pre-vaccination) and Day 43 (post-Dose 2/pre-vaccination)
Population: as for outcome 15
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | FLU-Q-PAN H7N9 Formulation 1_B Group | FLU-Q-PAN H7N9 Formulation 1_A Group | FLU-Q-PAN H7N9 Formulation 2_B Group | FLU-Q-PAN H7N9 Formulation 2_A Group | FLU-Q-PAN H7N9 Formulation 3_B Group | FLU-Q-PAN H7N9 Formulation 3_A Group | Placebo Group
Number analyzed (Participants) | 98 | 93 | 97 | 94 | 101 | 94 | 95
Ratio
  Day 22 | 1.1 [1.1 to 1.2] | 1.1 [1.1 to 1.2] | 1.3 [1.2 to 1.6] | 1.4 [1.2 to 1.6] | 1.5 [1.3 to 1.7] | 1.7 [1.4 to 2.1] | 1.0 [1.0 to 1.0]
  Day 43: number analyzed (Participants) | 96 | 83 | 85 | 83 | 89 | 84 | 82
  Day 43 | 2.7 [2.2 to 3.3] | 3.0 [2.4 to 3.6] | 2.7 [2.2 to 3.4] | 3.2 [2.6 to 3.9] | 2.6 [2.1 to 3.2] | 4.5 [3.5 to 5.7] | 1.0 [1.0 to 1.0]

20. Secondary Outcome: Anti-microneutralization (MN) Antibody Titers Against Vaccine-homologous H7N9 for a Subset of Participants
Description: Anti-MN antibody titers were expressed as GMTs. The GMTs calculations were performed by taking the antilog of the mean of the log titer transformations. Values for the neutralisation titers below the assay cut-off were assigned half the assay cut-off value for the purpose of GMT computation. MN analyses were performed on the MN subset that included approximately 420 participants (60 per group). The first 30 participants per treatment group were selected in the ≥65 age group and then the first 15 participants in 18 to 49 years and 50 to 64 years age groups. If there were not 15 participants for the 18 to 49 or 50 to 64 years age groups, they were selected whichever had the smaller number fully and then had a total of 30 for the total among these 2 age groups per treatment group. All samples were collected first, then selected for the subset.
Time Frame: At Day 1, Day 22 and Day 43
Population: Analysis was performed on the MN subset (selection of approximatively 50% participants from H7N9 vaccine groups and 50% participants from Placebo group) of the Per Protocol Set, which included all participants with no major protocol deviations that lead to exclusion at or prior to Day 43, who had data collected for MN at each visit and for whom immunogenicity data was available for the specified timepoints and specific assay.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | FLU-Q-PAN H7N9 Formulation 1_B Group | FLU-Q-PAN H7N9 Formulation 1_A Group | FLU-Q-PAN H7N9 Formulation 2_B Group | FLU-Q-PAN H7N9 Formulation 2_A Group | FLU-Q-PAN H7N9 Formulation 3_B Group | FLU-Q-PAN H7N9 Formulation 3_A Group | Placebo Group
Number analyzed (Participants) | 48 | 46 | 50 | 51 | 50 | 48 | 51
Titers
  Day 1 | 14.150 [NA to NA] — The Confidence Interval could not be calculated. | 14.150 [NA to NA] — The Confidence Interval could not be calculated. | 14.348 [14.0 to 14.8] | 14.150 [NA to NA] — The Confidence Interval could not be calculated. | 14.150 [NA to NA] — The Confidence Interval could not be calculated. | 14.356 [13.9 to 14.8] | 14.344 [14.0 to 14.7]
  Day 22 | 15.997 [14.3 to 17.8] | 15.724 [14.4 to 17.1] | 18.800 [14.7 to 24.1] | 17.232 [15.2 to 19.6] | 17.180 [14.8 to 19.9] | 18.218 [15.9 to 20.9] | 14.344 [14.0 to 14.7]
  Day 43: number analyzed (Participants) | 48 | 41 | 42 | 46 | 47 | 42 | 44
  Day 43 | 41.784 [31.4 to 55.6] | 42.453 [31.6 to 57.0] | 37.153 [27.5 to 50.2] | 40.926 [31.0 to 54.0] | 32.792 [25.9 to 41.5] | 54.297 [38.6 to 76.3] | 14.603 [14.0 to 15.3]

21. Secondary Outcome: Percentage of Seropositive Participants for Vaccine-homologous H7N9 MN Antibody Titers for a Subset of Participants
Description: A seropositive participant is a participant whose antibody titer was greater than or equal to the assay cut-off value.
  Note: The cut-off value for antibody titer was defined by the laboratory before the analysis. MN analyses were performed on the MN subset.
Time Frame: At Day 1, Day 22 and Day 43
Population: Analysis was performed on the MN subset (selection of approximatively 50% participants from H7N9 vaccine groups and 50% participants from Placebo group) of the Per Protocol Set, which included all participants with no major protocol deviations that lead to exclusion at or prior to Day 43, who had data for seropositivity of MN antibodies at each visit and for whom post-vaccination immunogenicity data was available for the specified timepoints and specific assay.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | FLU-Q-PAN H7N9 Formulation 1_B Group | FLU-Q-PAN H7N9 Formulation 1_A Group | FLU-Q-PAN H7N9 Formulation 2_B Group | FLU-Q-PAN H7N9 Formulation 2_A Group | FLU-Q-PAN H7N9 Formulation 3_B Group | FLU-Q-PAN H7N9 Formulation 3_A Group | Placebo Group
Number analyzed (Participants) | 48 | 46 | 50 | 51 | 50 | 48 | 51
Percentage of Participants
  Day 1 | 0 [0.0 to 7.4] | 0 [0.0 to 7.7] | 2.0 [0.1 to 10.6] | 0 [0.0 to 7.0] | 0 [0.0 to 7.1] | 2.1 [0.1 to 11.1] | 2.0 [0.0 to 10.4]
  Day 22 | 12.5 [4.7 to 25.2] | 13.0 [4.9 to 26.3] | 16.0 [7.2 to 29.1] | 19.6 [9.8 to 33.1] | 16 [7.2 to 29.1] | 25.0 [13.6 to 39.6] | 2.0 [0.0 to 10.4]
  Day 43: number analyzed (Participants) | 48 | 41 | 42 | 46 | 47 | 42 | 44
  Day 43 | 66.7 [51.6 to 79.6] | 73.2 [57.1 to 85.8] | 69.0 [52.9 to 82.4] | 67.4 [52.0 to 80.5] | 66.0 [50.7 to 79.1] | 76.2 [60.5 to 87.9] | 4.5 [0.6 to 15.5]

22. Secondary Outcome: Vaccine Response Rate (VRR) of Anti-MN Antibodies Against Vaccine-homologous H7N9 for a Subset of Participants
Description: VRR is expressed as the percentage of participants with a vaccine response defined as at least a 4-fold increase in antibody titer as compared to the antibody titer at Day 1 (pre-vaccination). Antibody titers below the cut-off of the assay were given an arbitrary value of half the cut-off for the purpose of vaccine response calculation. For VRR, the percentage of participants was calculated with Clopper-Pearson exact two-sided 95% CIs. MN analyses were performed on the MN subset.
Time Frame: At Day 22 and Day 43
Population: Analysis was performed on the MN subset (selection of approximatively 50% participants from H7N9 vaccine groups and 50% participants from Placebo group) of the Per Protocol Set, which included all participants with no major protocol deviations that lead to exclusion at or prior to Day 43, who had data for VRR at each visit and for whom post-vaccination immunogenicity data was available for the specified timepoints and specific assay.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | FLU-Q-PAN H7N9 Formulation 1_B Group | FLU-Q-PAN H7N9 Formulation 1_A Group | FLU-Q-PAN H7N9 Formulation 2_B Group | FLU-Q-PAN H7N9 Formulation 2_A Group | FLU-Q-PAN H7N9 Formulation 3_B Group | FLU-Q-PAN H7N9 Formulation 3_A Group | Placebo Group
Number analyzed (Participants) | 48 | 46 | 50 | 51 | 50 | 48 | 51
Percentage of Participants
  Day 22 | 2.1 [0.1 to 11.1] | 2.2 [0.1 to 11.5] | 8.0 [2.2 to 19.2] | 5.9 [1.2 to 16.2] | 6.0 [1.3 to 16.5] | 8.3 [2.3 to 20.0] | 0 [0.0 to 7.0]
  Day 43: number analyzed (Participants) | 48 | 41 | 42 | 46 | 47 | 42 | 44
  Day 43 | 45.8 [31.4 to 60.8] | 46.3 [30.7 to 62.6] | 38.1 [23.6 to 54.4] | 47.8 [32.9 to 63.1] | 34.0 [20.9 to 49.3] | 57.1 [41.0 to 72.3] | 0 [0.0 to 8.0]

ADVERSE EVENTS:
Time Frame: Solicited AEs: During the 7-day follow-up period after each vaccination. Unsolicited AEs: During the 21-day follow-up period after each vaccination. SAEs: From Day 1 up to Month 13.
Arm/Group | FLU-Q-PAN H7N9 Formulation 1_B Group | FLU-Q-PAN H7N9 Formulation 1_A Group | FLU-Q-PAN H7N9 Formulation 2_B Group | FLU-Q-PAN H7N9 Formulation 2_A Group | FLU-Q-PAN H7N9 Formulation 3_B Group | FLU-Q-PAN H7N9 Formulation 3_A Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/121 | 0/116 | 0/119 | 0/119 | 0/117 | 0/121 | 0/120
Serious Adverse Events (participants affected / at risk) | 3/121 | 3/116 | 10/119 | 4/119 | 6/117 | 5/121 | 7/120
Other Adverse Events (participants affected / at risk) | 40/121 | 32/116 | 33/119 | 34/119 | 30/117 | 39/121 | 33/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FLU-Q-PAN H7N9 Formulation 1_B Group (N=121) | FLU-Q-PAN H7N9 Formulation 1_A Group (N=116) | FLU-Q-PAN H7N9 Formulation 2_B Group (N=119) | FLU-Q-PAN H7N9 Formulation 2_A Group (N=119) | FLU-Q-PAN H7N9 Formulation 3_B Group (N=117) | FLU-Q-PAN H7N9 Formulation 3_A Group (N=121) | Placebo Group (N=120)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Right ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophagitis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Normal pressure hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic dissection (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FLU-Q-PAN H7N9 Formulation 1_B Group (N=121) | FLU-Q-PAN H7N9 Formulation 1_A Group (N=116) | FLU-Q-PAN H7N9 Formulation 2_B Group (N=119) | FLU-Q-PAN H7N9 Formulation 2_A Group (N=119) | FLU-Q-PAN H7N9 Formulation 3_B Group (N=117) | FLU-Q-PAN H7N9 Formulation 3_A Group (N=121) | Placebo Group (N=120)
Fatigue (General disorders) | 6 (21) | 5 (27) | 2 (6) | 2 (12) | 1 (6) | 3 (12) | 1 (9)
Injection site pain (General disorders) | 2 (6) | 4 (15) | 1 (3) | 2 (9) | 2 (9) | 2 (6) | 0 (0)
Chillis (General disorders) | 0 (0) | 0 (0) | 2 (6) | 1 (6) | 0 (0) | 3 (12) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 2 (6) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Pain (General disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (9) | 0 (0)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (3) | 1 (3)
Injection site swelling (General disorders) | 0 (0) | 2 (6) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Injection site warmth (General disorders) | 0 (0) | 1 (3) | 0 (0) | 1 (3) | 0 (0) | 1 (3) | 0 (0)
Injection site induration (General disorders) | 1 (6) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Administration site swelling (General disorders) | 0 (0) | 1 (3) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (3) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site haemorrhage (General disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (3) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Pyrexia (General disorders) | 0 (0) | 1 (3) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaccination site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foaming at mouth (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Hunger (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Injection site mass (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical device pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Suprapubic pain (General disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swelling face (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Thirst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Vessel puncture site pain (General disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (6) | 1 (3) | 3 (12) | 2 (12) | 3 (15) | 1 (3) | 7 (30)
Nausea (Gastrointestinal disorders) | 1 (6) | 1 (3) | 2 (9) | 2 (15) | 1 (3) | 2 (9) | 1 (6)
Abdominal pain (Gastrointestinal disorders) | 1 (6) | 0 (0) | 1 (3) | 1 (9) | 1 (3) | 1 (6) | 2 (9)
Constipation (Gastrointestinal disorders) | 2 (6) | 0 (0) | 1 (3) | 0 (0) | 2 (6) | 0 (0) | 1 (3)
Dyspepsia (Gastrointestinal disorders) | 1 (3) | 0 (0) | 1 (3) | 1 (3) | 0 (0) | 0 (0) | 2 (6)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0) | 1 (6) | 0 (0) | 1 (3) | 1 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (3) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (3) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Salivary gland enlargement (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tongue blistering (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (9) | 0 (0) | 2 (9) | 4 (15) | 0 (0) | 3 (9) | 1 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (12) | 0 (0) | 1 (3) | 2 (12) | 1 (3) | 2 (6) | 1 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 1 (3) | 3 (12) | 1 (3) | 1 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (9) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (3) | 2 (6)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 1 (3) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0) | 1 (3) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (6) | 0 (0) | 1 (3) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (3) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Muscle swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Headache (Nervous system disorders) | 5 (24) | 4 (24) | 3 (15) | 4 (18) | 2 (6) | 3 (12) | 3 (12)
Disturbance in attention (Nervous system disorders) | 1 (3) | 2 (6) | 1 (6) | 2 (6) | 2 (6) | 2 (6) | 1 (3)
Dizziness (Nervous system disorders) | 3 (9) | 3 (9) | 2 (6) | 2 (6) | 1 (3) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (3) | 0 (0) | 0 (0) | 1 (6) | 0 (0) | 2 (9) | 0 (0)
Migraine (Nervous system disorders) | 1 (6) | 0 (0) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 1 (3)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (6) | 1 (3)
Carotid arteriosclerosis (Nervous system disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parosmia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Tension headache (Nervous system disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (6) | 2 (6) | 3 (9) | 2 (6) | 2 (6) | 1 (3)
COVID-19 (Infections and infestations) | 1 (3) | 1 (3) | 3 (9) | 1 (3) | 0 (0) | 1 (3) | 1 (3)
Upper respiratory tract infection (Infections and infestations) | 2 (6) | 0 (0) | 1 (3) | 1 (3) | 0 (0) | 1 (3) | 1 (3)
Nasopharyngitis (Infections and infestations) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (3)
Bronchitis (Infections and infestations) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Localised infection (Infections and infestations) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Rhinitis (Infections and infestations) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (6)
Bacterial vaginosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Tinea pedis (Infections and infestations) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 2 (6) | 1 (6) | 1 (3) | 2 (6) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 0 (0) | 1 (6) | 0 (0) | 1 (3) | 2 (9)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3) | 0 (0) | 1 (3) | 2 (6) | 1 (3) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (3) | 1 (3) | 1 (3) | 1 (3) | 0 (0) | 1 (3) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (6) | 0 (0) | 0 (0) | 1 (3) | 1 (3) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Skin warm (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (6) | 2 (6) | 1 (3) | 1 (3) | 1 (3) | 1 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (6) | 1 (3) | 0 (0) | 1 (3) | 1 (3) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 1 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 1 (3) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (3) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (6) | 0 (0) | 1 (3) | 0 (0) | 2 (6) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (3) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 2 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (3) | 0 (0) | 1 (3) | 1 (3) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (3) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Corneal abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Heat exhaustion (Injury, poisoning and procedural complications) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Reactive gastropathy (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (3) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (3) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (9) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Blood urine present (Investigations) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymph node palpable (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Renal function test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Menstruation irregular (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostatic mass (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Testicular swelling (Reproductive system and breast disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine spasm (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (3) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Right ventricular failure (Cardiac disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (3) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 0 (0) | 0 (0)
Incontinence (Renal and urinary disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal cyst (Renal and urinary disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urge incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Deafness unilateral (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pruritus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral embolism (Vascular disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 2 (6) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-02-22): https://cdn.clinicaltrials.gov/large-docs/77/NCT04789577/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-17): https://cdn.clinicaltrials.gov/large-docs/77/NCT04789577/SAP_001.pdf